CLINICAL TRIAL: NCT01951625
Title: A Randomized Parallel-group, Placebo-controlled, Double-blind, Multi-center Dose Finding Phase II Trial Exploring the Pharmacodynamic Effects, Safety and Tolerability, and Pharmacokinetics of Four Dose Regimens of the Oral sGC Stimulator BAY1021189 Over 12 Weeks in Patients With Worsening Heart Failure With Reduced Ejection Fraction (HFrEF)
Brief Title: Phase IIb Safety and Efficacy Study of Four Dose Regimens of BAY1021189 in Patients With Heart Failure With Reduced Ejection Fraction Suffering From Worsening Chronic Heart Failure (SOCRATES-REDUCED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15371; 2013-002287-11 (EudraCT Number)
Record Dates: First submitted 2013-09-24; First posted 2013-09-26 (Estimated); Results first posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure
Keywords: Worsening Heart Failure; Heart Failure with Reduced Ejection Fraction
MeSH Terms: conditions — Heart Failure | interventions — vericiguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Vericiguat (BAY1021189) (10 mg) (Experimental): 2.5 mg orally once daily for 2 weeks, up-titration to 5 mg orally once daily for 2 weeks, up-titration to 10 mg orally once daily for 8 weeks
  Interventions: Drug: Vericiguat (BAY1021189) (1.25 mg); Drug: Vericiguat (BAY1021189) (5 mg)
- Vericiguat (BAY1021189) (5 mg) (Experimental): 2.5 mg orally once daily for 2 weeks, then 5 mg orally once daily for 10 weeks (with sham titration)
  Interventions: Drug: Vericiguat (BAY1021189) (1.25 mg); Drug: Vericiguat (BAY1021189) (5 mg)
- Vericiguat (BAY1021189) (2.5 mg) (Experimental): 2.5 mg orally once daily for 12 weeks (with sham titrations)
  Interventions: Drug: Vericiguat (BAY1021189) (1.25 mg)
- Vericiguat (BAY1021189) (1.25 mg) (Experimental): 1.25 mg orally once daily for 12 weeks (with sham titrations)
  Interventions: Drug: Vericiguat (BAY1021189) (1.25 mg)
- Placebo (Placebo Comparator): Orally once daily for 12 weeks (with sham titrations)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vericiguat (BAY1021189) (1.25 mg) — 1.25 mg BAY1021189 tablets
  Arms: Vericiguat (BAY1021189) (1.25 mg); Vericiguat (BAY1021189) (10 mg); Vericiguat (BAY1021189) (2.5 mg); Vericiguat (BAY1021189) (5 mg)
Drug: Vericiguat (BAY1021189) (5 mg) — 5 mg BAY1021189 tablets
  Arms: Vericiguat (BAY1021189) (10 mg); Vericiguat (BAY1021189) (5 mg)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Objective of the study is to find the optimal dose of the once daily oral soluble guanylate cyclase stimulator (sGC) BAY1021189 for Phase III that can be given in addition to standard therapy for heart failure with reduced ejection fraction (HFrEF).

ELIGIBILITY:
Inclusion Criteria:

* Worsening chronic heart failure (WCHF) requiring hospitalization (or intravenous diuretic treatment for HF without hospitalization) with initiation of study treatment after clinical stabilization
* Left ventricular ejection fraction (LVEF) <45% by echocardiography at randomization

Exclusion Criteria:

* Intravenous inotropes at any time after hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2013-11-29 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2015-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (142):
- United States (18):
  - Fountain Valley, California
  - Wilmington, Delaware
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Naples, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - New Orleans, Louisiana
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - Buffalo, New York
  - Columbus, Ohio
  - Fairfield, Ohio
  - Charleston, South Carolina
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Milwaukee, Wisconsin
- Australia (3):
  - Darlinghurst, New South Wales
  - Hobart, Tasmania
  - Prahran, Victoria
- Austria (5):
  - Sankt Pölten, Lower Austria
  - Graz, Styria
  - Linz, Upper Austria
  - Salzburg
  - Vienna
- Belgium (8):
  - Bruges
  - Bruxelles - Brussel
  - Ghent
  - Gilly
  - Huy
  - Mechelen
  - Mol
  - Roeselare
- Bulgaria (2):
  - Sofia
  - Stara Zagora
- Canada (5):
  - Toronto, Ontario
  - Montreal, Quebec
  - Saint-Jean-sur-Richelieu, Quebec
  - Sherbrooke, Quebec
  - Québec
- Czechia (5):
  - Hradec Králové
  - Kroměříž
  - Fakultni nemocnice Ostrava, Ostrava
  - Prague
  - Slaný
- Denmark (4):
  - Aalborg
  - Aarhus N
  - Hellerup
  - Viborg
- France (6):
  - Bron
  - La Tronche
  - Lille
  - Paris
  - Pessac
  - Rouen
- Germany (10):
  - München, Bavaria
  - Bad Homburg, Hesse
  - Frankfurt am Main, Hesse
  - Hanover, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Cologne, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Homburg, Saarland
  - Erfurt, Thuringia
  - Hamburg
- Greece (2):
  - Athens
  - Nea Ionia
- Hungary (3):
  - Budapest
  - Kistarcsa
  - Székesfehérvár
- Israel (9):
  - Afula
  - Ashkelon
  - Hadera
  - Jerusalem
  - Petah Tikva
  - Rehovot
  - Tel Aviv
  - Tiberias
  - Zrifin
- Italy (8):
  - Bergamo, Lombardy
  - Brescia, Lombardy
  - Como, Lombardy
  - Milan, Lombardy
  - Pavia, Lombardy
  - Ancona, The Marches
  - Arezzo, Tuscany
  - Verona, Veneto
- Japan (20):
  - Iizuka, Fukuoka
  - Himeji, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Sendai, Miyagi
  - Naha, Okinawa
  - Takatsuki, Osaka
  - Yao, Osaka
  - Ureshino, Saga-ken
  - Komatsushimachō, Tokushima
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Fukui
  - Hiroshima
  - Kumamoto
  - Nagasaki
  - Tokushima
  - Toyama
- Netherlands (5):
  - Amsterdam
  - Deventer
  - Heerenveen
  - Leeuwarden
  - Veldhoven
- Poland (7):
  - Bialystok
  - Krakow
  - Legnica
  - Lodz
  - Olsztyn
  - Poznan
  - Warsaw
- Singapore, Singapore
- Seoul, South Korea
- Spain (5):
  - L'Hospitalet de Llobregat, Barcelona
  - Santander, Cantabria
  - Majadahonda, Madrid
  - Barcelona
  - Valencia
- Sweden (6):
  - Helsingborg
  - Karlstad
  - Linköping
  - Malmo
  - Örebro
  - Stockholm
- Switzerland (4):
  - Liestal, Basel-Landschaft
  - Bruderholz
  - Lugano
  - Zurich
- Taiwan (3):
  - Kaohsiung City
  - New Taipei City
  - Taipei
- United Kingdom (2):
  - Chesterfield, Derbyshire
  - Stevenage, Hertfordshire

REFERENCES:
- [Result] Pieske B, Butler J, Filippatos G, Lam C, Maggioni AP, Ponikowski P, Shah S, Solomon S, Kraigher-Krainer E, Samano ET, Scalise AV, Muller K, Roessig L, Gheorghiade M; SOCRATES Investigators and Coordinators. Rationale and design of the SOluble guanylate Cyclase stimulatoR in heArT failurE Studies (SOCRATES). Eur J Heart Fail. 2014 Sep;16(9):1026-38. doi: 10.1002/ejhf.135. Epub 2014 Jul 24. PMID 25056511
- [Result] Gheorghiade M, Greene SJ, Butler J, Filippatos G, Lam CS, Maggioni AP, Ponikowski P, Shah SJ, Solomon SD, Kraigher-Krainer E, Samano ET, Muller K, Roessig L, Pieske B; SOCRATES-REDUCED Investigators and Coordinators. Effect of Vericiguat, a Soluble Guanylate Cyclase Stimulator, on Natriuretic Peptide Levels in Patients With Worsening Chronic Heart Failure and Reduced Ejection Fraction: The SOCRATES-REDUCED Randomized Trial. JAMA. 2015 Dec 1;314(21):2251-62. doi: 10.1001/jama.2015.15734. PMID 26547357
- [Derived] Ruehs H, Klein D, Frei M, Grevel J, Austin R, Becker C, Roessig L, Pieske B, Garmann D, Meyer M. Population Pharmacokinetics and Pharmacodynamics of Vericiguat in Patients with Heart Failure and Reduced Ejection Fraction. Clin Pharmacokinet. 2021 Nov;60(11):1407-1421. doi: 10.1007/s40262-021-01024-y. Epub 2021 Jun 4. PMID 34086190
- [Derived] Kramer F, Voss S, Roessig L, Igl BW, Butler J, Lam CSP, Maggioni AP, Shah SJ, Pieske B. Evaluation of high-sensitivity C-reactive protein and uric acid in vericiguat-treated patients with heart failure with reduced ejection fraction. Eur J Heart Fail. 2020 Sep;22(9):1675-1683. doi: 10.1002/ejhf.1787. Epub 2020 Mar 25. PMID 32216011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 144 centers in 24 countries between 29 November 2013 (first subject first visit) and 09 June 2015 (last subject last visit).
Pre-assignment Details: Overall 632 subjects were enrolled, of them 176 were screen failure and 456 were randomized. One subject did not receive study drug after randomization. Among the 455 subjects who received study drug 348 completed the study (that is completed both the treatment and follow-up periods) and 108 subjects did not complete the study.
Groups:
- Placebo: Subjects received placebo matched to vericiguat (Verquvo, BAY1021189) orally once daily for 12 weeks. Sham titrations included on Days 14 and 28.
- BAY1021189 1.25 Milligram (mg): Subjects received vericiguat (Verquvo, BAY1021189) 1.25 mg orally once daily for 12 weeks. Sham titrations included on Days 14 and 28.
- BAY1021189 2.5 mg: Subjects received vericiguat (Verquvo, BAY1021189) 2.5 mg orally once daily for 12 weeks. Sham titrations included on Days 14 and 28.
- BAY1021189 From 2.5 to 5 mg: Subjects received vericiguat (Verquvo, BAY1021189) for 12 weeks, starting on 2.5 mg once daily with potential up-titration to 5 mg once daily after 14 or 28 days. Sham titration included on Day 28.
- BAY1021189 From 2.5 to 10 mg: Subjects received vericiguat (Verquvo, BAY1021189) for 12 weeks, starting on 2.5 mg once daily with potential up-titration to 5 mg once daily after 14 days, and up-titration to 10 mg once daily after 28 days.
Period: Treatment Period
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Started | 92 | 91 | 91 | 91 | 91
Completed | 73 | 70 | 76 | 69 | 74
Not Completed | 19 | 21 | 15 | 22 | 17
Not completed — Protocol Violation | 2 | 0 | 1 | 3 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Protocol driven decision point | 0 | 5 | 0 | 2 | 1
Not completed — Non compliance with study drug | 1 | 2 | 2 | 0 | 0
Not completed — Death | 3 | 2 | 2 | 1 | 2
Not completed — Adverse Event | 7 | 10 | 9 | 8 | 8
Not completed — Withdrawal by Subject | 5 | 2 | 1 | 7 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0
Period: Follow Up Period
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Started | 87 | 88 | 88 | 87 | 88
Completed | 79 | 79 | 84 | 76 | 78
Not Completed | 8 | 9 | 4 | 11 | 10
Not completed — Non-compliance with study drug | 1 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 3 | 2 | 2 | 1
Not completed — Logistical difficulties | 1 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 2 | 3 | 5
Not completed — Withdrawal by Subject | 4 | 1 | 0 | 5 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg | Total
Number analyzed (Participants) | 92 | 91 | 91 | 91 | 91 | 456
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (13.1) | 67.6 (12.9) | 67.6 (11.5) | 66.7 (11.6) | 68.9 (12.4) | 67.6 (12.3)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 38 | 38 | 30 | 38 | 28 | 172
  65-75 | 26 | 19 | 37 | 32 | 34 | 148
  > 75 | 28 | 34 | 24 | 21 | 29 | 136
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 19 | 17 | 14 | 90
  Male | 73 | 70 | 72 | 74 | 77 | 366

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Log-Transformed N-Terminal Pro-Brain Natriuretic Peptide (NTproBNP) to Week 12
Description: Log-Transformed N-Terminal Pro-Brain Natriuretic Peptide (NTproBNP) is a circulating plasma biomarker of cardiovascular function and prognosis in heart failure.
Time Frame: Baseline, Week 12
Population: Per Protocol Set (PPS)
Measure: Mean (Standard Deviation); unit: log-transformed picograms per milliliter
Groups:
- Pooled 2.5 mg up to 10 mg: The three highest dose arms (BAY1021189 2.5 mg, 2.5-5 mg, and 2.5-10 mg) were pooled.
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg | Pooled 2.5 mg up to 10 mg
Number analyzed (Participants) | 69 | 69 | 73 | 67 | 73 | 213
log-transformed picograms per milliliter | -0.28 (0.8197) | -0.265 (0.7658) | -0.32 (0.7799) | -0.353 (0.8404) | -0.529 (0.9475) | -0.402 (0.8603)
Statistical Analysis 1: Comparison: Placebo vs Pooled 2.5 mg up to 10 mg; For the primary analysis, the three highest active treatment groups (BAY1021189 2.5mg, BAY1021189 2.5 to 5mg, BAY1021189 2.5 to 10mg) were pooled and compared to the assigned placebo treatment group with a one-sided two-sample t-test at the significance level of 5 percent (%). Results are reported including 90% confidence intervals (CI) for the difference of means. The difference between the pooled treatment group and the placebo group is difference of means on the log scale; Test type: Other; p = 0.1506, t-test, 1 sided; Log-Scale mean difference = -0.122, 90% CI 2-sided [-0.32 to 0.07]
Statistical Analysis 2: Comparison: Placebo vs BAY1021189 From 2.5 to 10 mg; In case of a significant result in the primary analysis of the primary endpoint, pairwise comparisons to Placebo were performed in a hierarchical manner (from BAY1021189 from 2.5 to 10mg dose arm to BAY1021189 1.25mg dose arm). In case of non-significance of the primary analyses, these secondary analyses were specified as exploratory only, since the primary analyses were not significant; Test type: Other; p = 0.0483, t-test, 1 sided; Log-Scale mean difference = -0.2494, 90% CI 2-sided [-0.5 to 0]
Statistical Analysis 3: Comparison: Placebo vs BAY1021189 From 2.5 to 5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.3042, t-test, 1 sided; Log-Scale mean difference = -0.0731, 90% CI 2-sided [-0.31 to 0.16]
Statistical Analysis 4: Comparison: Placebo vs BAY1021189 2.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.3841, t-test, 1 sided; Log-Scale mean difference = -0.0396, 90% CI 2-sided [-0.26 to 0.18]
Statistical Analysis 5: Comparison: Placebo vs BAY1021189 1.25 Milligram (mg); In case of a significant result in the primary analysis of the primary endpoint, pairwise comparisons to Placebo were performed in a hierarchical manner (from BAY1021189 from 2.5 to 10mg dose arm to BAY1021189 1.25mg dose arm). In case of non-significance of the primary analyses, these secondary analyses were specified as exploratory only; Test type: Other; p = 0.5444, t-test, 1 sided; Log-Scale mean difference = 0.0151, 90% CI 2-sided [-0.21 to 0.24]

2. Other Pre Specified Outcome: Changes in Heart Function as Measured by Echocardiography, Left Ventricular End-Diastolic Volume (LVEDV), and Left Ventricular End-Systolic Volume (LVESV) From Baseline to Week 12
Description: Left Ventricular End-Diastolic Volume (LVEDV) and Left ventricular end-systolic volume (LVESV) are measured echocardiography parameter. These are acquired during a non-invasive echocardiography examination.
Time Frame: Baseline, Week 12
Population: Evaluable subjects in full analysis set (FAS).
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 92 | 91 | 91 | 91 | 91
milliliter
  Change in LVEDV: number analyzed (Participants) | 70 | 65 | 69 | 63 | 70
  Change in LVEDV | -7.259 (40.676) | -5.525 (34.75) | -9.632 (35.081) | -17.093 (53.307) | -7.324 (31.896)
  Change in LVESV: number analyzed (Participants) | 70 | 65 | 69 | 63 | 71
  Change in LVESV | -6.83 (32.407) | -8.585 (27.385) | -10.935 (27.146) | -15.485 (43.191) | -11.017 (26.525)

3. Other Pre Specified Outcome: Changes in Heart Function as Measured by Echocardiography, Left Ventricular Ejection Fraction (LVEF), From Baseline to Week 12
Description: The left ventricular ejection fraction work index (LVEF) is a calculated echocardiography parameter. LVEF is derived from the directly measured parameters left ventricular end-diastolic volume (LVEDV) and left ventricular end-systolic volume (LVESV). These 2 parameters are acquired during a noninvasive echocardiography examination. Formula: LVEF = 100*(LVEDV - LVESV)/LVEDV.
Time Frame: Baseline, Week 12
Population: Evaluable subjects in full analysis set (FAS).
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 92 | 91 | 91 | 91 | 91
percentage | 1.515 (4.736) | 2.84 (3.635) | 2.741 (4.371) | 2.07 (4.808) | 3.682 (6.19)

4. Other Pre Specified Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure to Week 12
Description: Blood pressure was measured by monitor measurements after 10 minutes resting in a supine position (3 measurements taken approximately 2 minutes apart).The changes in blood pressure were recorded and the mean of the three measurements was analyzed.
Time Frame: Baseline, Week 12
Population: Evaluable subjects in safety analysis set (SAF).
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 92 | 91 | 90 | 91 | 91
millimeter of mercury (mmHg)
  Change in SBP: number analyzed (Participants) | 73 | 70 | 75 | 69 | 74
  Change in SBP | -5.142 (12.829) | -4.033 (13.3) | -3.733 (16.509) | -3.043 (15.934) | -5.64 (15.509)
  Change in DBP: number analyzed (Participants) | 73 | 70 | 75 | 69 | 74
  Change in DBP | -4.173 (8.6) | -0.486 (9.298) | -2.938 (11.101) | -1.338 (9.528) | -4.045 (10.604)

5. Other Pre Specified Outcome: Change From Baseline in Heart Rate to Week 12
Description: Heart rate was measured after 10 minutes resting in a supine position (3 measurements taken approximately 2 minutes apart). The changes in heart rate were recorded and the mean of the three measurements was analyzed.
Time Frame: Baseline, Week 12
Population: Evaluable subjects in safety analysis set (SAF).
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 92 | 91 | 90 | 91 | 91
Beats per minute | -0.562 (12.897) | -0.352 (10.153) | -1.556 (10.2) | -0.99 (11.295) | 0.545 (10.636)

6. Other Pre Specified Outcome: Number of Subjects With Clinical Events (Heart Failure [HF] Hospitalization and Cardio-Vascular [CV] Mortality)
Description: Clinical events (heart failure and mortality) were analyzed as CV death, and HF hospitalization at specified time points.
Time Frame: Baseline until 16 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 92 | 91 | 91 | 91 | 91
Participants
  HF hospitalizations | 21 | 18 | 20 | 10 | 9
  CV death | 6 | 5 | 4 | 2 | 4

7. Other Pre Specified Outcome: Number of Subjects With Implantable Cardioverter Defibrillators Cardiac Resynchronization Therapy With Defibrillation (ICD/CRT-D) Therapy
Description: ICD / CRT with defibrillation therapy (CRT-D) included previous appropriate interventions such as shocks or anti-tachycardic pacing (ATP) when diagnostic of sustained ventricular tachycardias in pre defined rapid zone.
Time Frame: Baseline upto 16 weeks
Population: No analysis was performed for this end point.
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Other Pre Specified Outcome: Number of Subjects With Treatment-Emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a subject who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; and another medically important serious event as judged by the investigator. AEs are considered to be treatment-emergent if they have started or worsened after first application of study drug up to 5 days after end of treatment with study drug.
Time Frame: From the start of study treatment upto 5 days after the last dose of study drug
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 92 | 91 | 90 | 91 | 91
Participants | 66 | 60 | 62 | 62 | 56

9. Other Pre Specified Outcome: Change in Biomarkers From Baseline to Week 12: Osteopontin (ng/mL)
Time Frame: Baseline, Week 12
Population: Evaluable subjects in FAS
Measure: Mean (Standard Deviation); unit: nanogram(s)/milliliter (ng/mL)
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 73 | 69 | 73 | 65 | 71
nanogram(s)/milliliter (ng/mL) | 2.79 (42.049) [lower limit 42.049] | 3.812 (39.248) [lower limit 39.248] | 3.266 (52.957) [lower limit 52.957] | 8.485 (41.97) [lower limit 41.97] | 3.709 (36.048) [lower limit 36.048]

10. Other Pre Specified Outcome: Change in Biomarkers From Baseline to Week 12: TIMP-4 (pg/mL)
Description: TIMP-4: tissue inhibitor of matrix metalloproteinases 4
Time Frame: Baseline, Week 12
Population: Evaluable subjects in FAS
Measure: Mean (Standard Deviation); unit: picogram(s)/millilitre (pg/mL)
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 73 | 69 | 72 | 67 | 72
picogram(s)/millilitre (pg/mL) | 451.889 (1392.03) [lower limit 1392.03] | 1128.635 (1949.351) [lower limit 1949.351] | 643.626 (1441.954) [lower limit 1441.954] | 876.584 (1559.768) [lower limit 1559.768] | 397.603 (1420.223) [lower limit 1420.223]

11. Other Pre Specified Outcome: Change in Biomarkers From Baseline to Week 12: cGMP (Pmol/mL)
Description: cGMP: cyclic guanosine monophosphate
Time Frame: Baseline, Week 12
Population: Evaluable subjects in FAS
Measure: Mean (Standard Deviation); unit: picomole(s)/milliliter (pmol/mL)
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 73 | 69 | 73 | 66 | 71
picomole(s)/milliliter (pmol/mL) | 78.874 (143.321) [lower limit 143.321] | 79.767 (123.031) [lower limit 123.031] | 92.352 (121.477) [lower limit 121.477] | 80.888 (114.09) [lower limit 114.09] | 63.563 (127.448) [lower limit 127.448]

12. Other Pre Specified Outcome: Change in Biomarkers From Baseline to Week 12: PIIINP (mcg/L)
Description: PIIINP: pro-collagen III N-terminal peptide
Time Frame: Baseline, Week 12
Population: Evaluable subjects in FAS
Measure: Mean (Standard Deviation); unit: microgram(s)/liter (mcg/L)
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 70 | 69 | 72 | 67 | 73
microgram(s)/liter (mcg/L) | -0.701 (7.246) [lower limit 7.246] | 0.092 (3.958) [lower limit 3.958] | 0.106 (5.145) [lower limit 5.145] | -0.71 (3.774) [lower limit 3.774] | -0.321 (4.452) [lower limit 4.452]

13. Other Pre Specified Outcome: Change in Biomarkers From Baseline to Week 12: GDF-15 (pg/mL)
Description: GDF-15: growth differentiation factor 15
Time Frame: Baseline, Week 12
Population: Evaluable subjects in FAS
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 73 | 69 | 73 | 66 | 71
pg/mL | 429.432 (3212.229) [lower limit 3212.229] | 496.456 (3132.738) [lower limit 3132.738] | 285.472 (2837.237) [lower limit 2837.237] | 468.369 (1786.062) [lower limit 1786.062] | 244.63 (2906.763) [lower limit 2906.763]

14. Other Pre Specified Outcome: Change in Biomarkers From Baseline to Week 12: ST2 (pg/mL)
Description: ST2: suppression of tumorigenicity 2
Time Frame: Baseline, Week 12
Population: Evaluable subjects in FAS
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 73 | 69 | 72 | 67 | 72
pg/mL | 9457.677 (54702.45) [lower limit 54702.45] | 1623.869 (25086.72) [lower limit 25086.72] | -1217.77 (35166.41) [lower limit 35166.41] | 6933.941 (20747.71) [lower limit 20747.71] | 3681.668 (32293.77) [lower limit 32293.77]

15. Other Pre Specified Outcome: Change in Biomarkers From Baseline to Week 12: Gal-3 (μg/mL)
Description: Gal-3: Galectin-3
Time Frame: Baseline, Week 12
Population: Evaluable subjects in FAS
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
Number analyzed (Participants) | 72 | 68 | 73 | 64 | 71
mcg/L | 0.802 (13.818) [lower limit 13.818] | 0.233 (6.208) [lower limit 6.208] | -0.287 (3.729) [lower limit 3.729] | 0.064 (5.64) [lower limit 5.64] | -0.38 (4.551) [lower limit 4.551]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs were collected after first application of study medication up to 5 calendar days after end of treatment with study medication.
Arm/Group | Placebo | BAY1021189 1.25 Milligram (mg) | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
All-Cause Mortality (participants affected / at risk) | 6/92 | 6/91 | 5/90 | 3/91 | 4/91
Serious Adverse Events (participants affected / at risk) | 30/92 | 26/91 | 26/90 | 20/91 | 25/91
Other Adverse Events (participants affected / at risk) | 24/92 | 25/91 | 20/90 | 23/91 | 28/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=92) | BAY1021189 1.25 Milligram (mg) (N=91) | BAY1021189 2.5 mg (N=90) | BAY1021189 From 2.5 to 5 mg (N=91) | BAY1021189 From 2.5 to 10 mg (N=91)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 8 (14) | 13 (14) | 10 (11) | 3 (4) | 3 (4)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 5 (5) | 2 (3) | 5 (5) | 3 (6) | 4 (4)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (3) | 3 (3) | 2 (2) | 3 (4)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transplant evaluation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 4 (4) | 2 (2) | 1 (1) | 3 (3)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter placement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=92) | BAY1021189 1.25 Milligram (mg) (N=91) | BAY1021189 2.5 mg (N=90) | BAY1021189 From 2.5 to 5 mg (N=91) | BAY1021189 From 2.5 to 10 mg (N=91)
Cardiac failure chronic (Cardiac disorders) | 4 (5) | 1 (1) | 5 (5) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 5 (6) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (7)
Nausea (Gastrointestinal disorders) | 3 (4) | 5 (6) | 3 (3) | 1 (1) | 1 (1)
Asthenia (General disorders) | 3 (3) | 0 (0) | 2 (2) | 5 (5) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 2 (2) | 2 (2) | 5 (6)
Dizziness (Nervous system disorders) | 5 (6) | 3 (3) | 2 (2) | 2 (2) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 3 (3) | 2 (3) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 8 (8) | 4 (4) | 4 (4) | 4 (4)
Hypotension (Vascular disorders) | 6 (6) | 5 (5) | 5 (6) | 4 (4) | 14 (17)

LIMITATIONS AND CAVEATS:
Endpoints of "Change in 'health-related quality of life', 'Composite Congestion Score', 'NYHA function class', and 'background heart failure therapies' were assessed as exploratory. "Incidence of atrial fibrillation" is reported in AE summary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No